CLINICAL TRIAL: NCT00832442
Title: Collaborative Systematic Overview of Randomised Controlled Trials of Beta-Blockers in the Treatment of Heart Failure
Acronym: BB-META-HF
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: CTEU08/d5/BBHF
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2009-01

CONDITIONS: Heart Failure
Keywords: Beta blocker; Heart Failure; Meta analysis; Individual patient data
MeSH Terms: conditions — Heart Failure | interventions — Adrenergic beta-Antagonists; Metoprolol; bucindolol; Carvedilol; Bisoprolol; Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Beta blocker
  Interventions: Drug: Beta blocker
- Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Beta blocker — as determined by individual study
  Other Names: Metoprolol; Bucindolol; Carvedilol; Bisoprolol; Nebivolol
  Groups: Beta blocker
Other: Placebo — in addition to usual care
  Groups: Placebo

SUMMARY:
Several large trials have shown that beta-blocker treatment reduces the risk of death and hospital admission in patients with symptomatic heart failure. Unfortunately, survey data suggests relatively poor utilisation of beta-blockers, despite ample evidence for good tolerability. Additionally there are several important unanswered questions, such as clinical efficacy for specific sub-populations (women, the elderly and patients with diabetes or other co-morbidities) and the effect of beta-blockers in combination with other medications. Previous meta-analyses, based on published tabular data, have been conducted although this approach has important biases and limitations.

We plan to perform a carefully conducted systematic review of individual patient data from the major randomised trials of beta-blockers in heart failure. The goals of this collaborative project are to clarify the overall efficacy of beta-blockers and identify sub-groups that show particular benefit, thereby increasing the use of beta-blockers, reducing adverse clinical outcomes and the high costs associated with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Randomised control trials of beta-blocker versus control in patients with documented heart failure
* Unconfounded trials only (in which one treatment group differed from another only by the beta-blocker therapy of interest)
* Randomization process precluded prior knowledge of the next treatment (for example trials in which treatment allocation was alternate or based on odd or even dates would not be included)

Exclusion Criteria:

* Trial sample size of less than 300 patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Meta-Analysis of randomised controlled trials investigating mortality & morbidity of placebo versus beta-blockers in heart failure
Sampling Method: Non-Probability Sample
Enrollment: 18240 (Estimated)
Dates: Start 2008-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Beta-blocker therapy improves overall mortality and morbidity in symptomatic heart failure in an individual patient meta-analysis | variable (time to event)

SECONDARY OUTCOMES:
Beta-blocker therapy improves mortality and morbidity in both elderly patients and women | variable (time to event)
Beta-blocker therapy improves mortality and morbidity in patients with co-morbidities (diabetes, renal dysfunction, COPD, peripheral arterial disease or atrial fibrillation) | variable (time to event)
The benefit of beta-blockers is not modified by concomitant cardiovascular therapy | variable (time to event)
The benefit of beta-blockers is independent of left ventricular ejection fraction at baseline | variable (time to event)
The clinical benefit is dependent on the resting heart rate achieved whatever the dose achieved or agent used | variable (time to event)
Adverse side effects of beta blocker therapy do not significantly impact on clinical benefit (as a whole and in relevant sub-groups) | variable (time to event)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Flather, Study Chair — Royal Brompton Hospital, London; Luis Manzano, Study Chair — Universidad de Alcala, Madrid; Dipak Kotecha, Study Chair — Royal Brompton Hospital, London; Henry Krum, Study Chair — Monash University, Melbourne
Locations (2):
- United Kingdom (2):
  - Clinical Trials & Evaluation Unit, Royal Brompton Hospital, London
  - Centre for Statistics in Medicine, University of Oxford, Oxford

REFERENCES:
- [Background] Waagstein F, Bristow MR, Swedberg K, Camerini F, Fowler MB, Silver MA, Gilbert EM, Johnson MR, Goss FG, Hjalmarson A. Beneficial effects of metoprolol in idiopathic dilated cardiomyopathy. Metoprolol in Dilated Cardiomyopathy (MDC) Trial Study Group. Lancet. 1993 Dec 11;342(8885):1441-6. doi: 10.1016/0140-6736(93)92930-r. PMID 7902479
- [Background] A randomized trial of beta-blockade in heart failure. The Cardiac Insufficiency Bisoprolol Study (CIBIS). CIBIS Investigators and Committees. Circulation. 1994 Oct;90(4):1765-73. doi: 10.1161/01.cir.90.4.1765. PMID 7923660
- [Background] Randomised, placebo-controlled trial of carvedilol in patients with congestive heart failure due to ischaemic heart disease. Australia/New Zealand Heart Failure Research Collaborative Group. Lancet. 1997 Feb 8;349(9049):375-80. PMID 9033462
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] The Cardiac Insufficiency Bisoprolol Study II (CIBIS-II): a randomised trial. Lancet. 1999 Jan 2;353(9146):9-13. PMID 10023943
- [Background] Packer M, Coats AJ, Fowler MB, Katus HA, Krum H, Mohacsi P, Rouleau JL, Tendera M, Castaigne A, Roecker EB, Schultz MK, DeMets DL; Carvedilol Prospective Randomized Cumulative Survival Study Group. Effect of carvedilol on survival in severe chronic heart failure. N Engl J Med. 2001 May 31;344(22):1651-8. doi: 10.1056/NEJM200105313442201. PMID 11386263
- [Background] Beta-Blocker Evaluation of Survival Trial Investigators; Eichhorn EJ, Domanski MJ, Krause-Steinrauf H, Bristow MR, Lavori PW. A trial of the beta-blocker bucindolol in patients with advanced chronic heart failure. N Engl J Med. 2001 May 31;344(22):1659-67. doi: 10.1056/NEJM200105313442202. PMID 11386264
- [Background] Flather MD, Shibata MC, Coats AJ, Van Veldhuisen DJ, Parkhomenko A, Borbola J, Cohen-Solal A, Dumitrascu D, Ferrari R, Lechat P, Soler-Soler J, Tavazzi L, Spinarova L, Toman J, Bohm M, Anker SD, Thompson SG, Poole-Wilson PA; SENIORS Investigators. Randomized trial to determine the effect of nebivolol on mortality and cardiovascular hospital admission in elderly patients with heart failure (SENIORS). Eur Heart J. 2005 Feb;26(3):215-25. doi: 10.1093/eurheartj/ehi115. Epub 2005 Jan 9. PMID 15642700
- [Background] Dargie HJ. Effect of carvedilol on outcome after myocardial infarction in patients with left-ventricular dysfunction: the CAPRICORN randomised trial. Lancet. 2001 May 5;357(9266):1385-90. doi: 10.1016/s0140-6736(00)04560-8. PMID 11356434
- [Derived] Banerjee A, Pasea L, Chung SC, Direk K, Asselbergs FW, Grobbee DE, Kotecha D, Anker SD, Dyszynski T, Tyl B, Denaxas S, Lumbers RT, Hemingway H. A population-based study of 92 clinically recognized risk factors for heart failure: co-occurrence, prognosis and preventive potential. Eur J Heart Fail. 2022 Mar;24(3):466-480. doi: 10.1002/ejhf.2417. Epub 2022 Jan 26. PMID 34969173
- [Derived] Karwath A, Bunting KV, Gill SK, Tica O, Pendleton S, Aziz F, Barsky AD, Chernbumroong S, Duan J, Mobley AR, Cardoso VR, Slater K, Williams JA, Bruce EJ, Wang X, Flather MD, Coats AJS, Gkoutos GV, Kotecha D; card AIc group and the Beta-blockers in Heart Failure Collaborative Group. Redefining beta-blocker response in heart failure patients with sinus rhythm and atrial fibrillation: a machine learning cluster analysis. Lancet. 2021 Oct 16;398(10309):1427-1435. doi: 10.1016/S0140-6736(21)01638-X. Epub 2021 Aug 30. PMID 34474011
- [Derived] Kotecha D, Manzano L, Krum H, Rosano G, Holmes J, Altman DG, Collins PD, Packer M, Wikstrand J, Coats AJ, Cleland JG, Kirchhof P, von Lueder TG, Rigby AS, Andersson B, Lip GY, van Veldhuisen DJ, Shibata MC, Wedel H, Bohm M, Flather MD; Beta-Blockers in Heart Failure Collaborative Group. Effect of age and sex on efficacy and tolerability of beta blockers in patients with heart failure with reduced ejection fraction: individual patient data meta-analysis. BMJ. 2016 Apr 20;353:i1855. doi: 10.1136/bmj.i1855. PMID 27098105
- [Derived] Kotecha D, Holmes J, Krum H, Altman DG, Manzano L, Cleland JG, Lip GY, Coats AJ, Andersson B, Kirchhof P, von Lueder TG, Wedel H, Rosano G, Shibata MC, Rigby A, Flather MD; Beta-Blockers in Heart Failure Collaborative Group. Efficacy of beta blockers in patients with heart failure plus atrial fibrillation: an individual-patient data meta-analysis. Lancet. 2014 Dec 20;384(9961):2235-43. doi: 10.1016/S0140-6736(14)61373-8. Epub 2014 Sep 2. PMID 25193873
- [Derived] Kotecha D, Manzano L, Altman DG, Krum H, Erdem G, Williams N, Flather MD; Beta-Blockers in Heart Failure Collaborative Group. Individual patient data meta-analysis of beta-blockers in heart failure: rationale and design. Syst Rev. 2013 Jan 18;2:7. doi: 10.1186/2046-4053-2-7. PMID 23327629
- See also: Monash Centre of Cardiovascular Research & Education (CCRE) in Therapeutics — http://www.ccretherapeutics.org.au/